CLINICAL TRIAL: NCT00004763
Title: Phase II Randomized Study of Leuprolide Vs Oral Contraceptive Therapy Vs Leuprolide and Oral Contraceptive Therapy for Ovarian Hyperandrogenism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Baylor College of Medicine (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/11717; BCM-11717
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Hyperandrogenism
Keywords: endocrine disorders; hyperandrogenism; rare disease
MeSH Terms: conditions — Hyperandrogenism; Endocrine System Diseases; Rare Diseases | interventions — Leuprolide; ovcon 35

INTERVENTIONS:
Drug: leuprolide
Drug: Ethinyl estradiol/norethindrone

SUMMARY:
OBJECTIVES:

I. Evaluate the beneficial effects of leuprolide depot, oral contraceptive therapy, and leuprolide/oral contraceptive therapy in the management of patients with ovarian hyperandrogenism.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are randomly assigned to a 6-month course of leuprolide versus ethinyl estradiol/norethindrone (Ovcon 35) versus leuprolide plus Ovcon 35. Leuprolide is administered intramuscularly in depot form every 28 days.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Disease Characteristics

* Ovarian hyperandrogenism with Lorenzo hirsutism score 7 to 20, with or without severe acne
* Serum hormone levels: Follicle-stimulating hormone no greater than 40 mIU/mL Luteinizing hormone no greater than 40 mIU/mL Testosterone 60 to 200 ng/dL Dehydroepiandrosterone sulfate no greater than 430 micrograms/dL 17-hydroxyprogesterone no greater than 3.3 ng/mL in follicular phase Prolactin no greater than 18 ng/dL
* No adrenal or ovarian tumors

Prior/Concurrent Therapy

* At least 6 months since exogenous steroids At least 48 hours since drugs other than acetaminophen, ibuprofen, and aspirin

Patient Characteristics

* No malignancy, including the following carcinomas: Breast Cervix Ovary Uterus No other serious illness No cigarette smokers No nursing women No pregnancy within 6 months prior to entry

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45
Dates: Start 1993-01

CONTACTS AND LOCATIONS:
Overall Officials: Karen E. Elkind-Hirsch, Study Chair — Baylor College of Medicine